CLINICAL TRIAL: NCT05593978
Title: Culinary Medicine to Enhance Protein Intake on Muscle Quality in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Muscle Culinary Medicine
Record Dates: First submitted 2022-02-07; First posted 2022-10-26 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Sarcopenia
Keywords: Culinary medicine; muscle synthesis; muscle strength; protein intake
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culinary Medicine (Experimental): Those in this group will receive culinary medicine, which includes cooking videos and educational videos to help educate on ways to increase protein intake through lean ground beef.
  Interventions: Behavioral: Culinary Medicine
- Control (Other): This group will only receive recipes containing lean ground beef to help increase protein intake.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Culinary Medicine — The CM-group will receive weekly cooking demonstrations and education videos via electronic links for 16 weeks, and three nutrition education based on the content of the Nutrition Care Manual from the Academy of Nutrition and Dietetics to show age-appropriate recipes with correct preparation methods and different cooking methods for lean ground red meat to increase protein consumption.
  Arms: Culinary Medicine
Behavioral: Control — The CN-group will receive weekly recipes via electronic links without the culinary medicine intervention.
  Arms: Control

SUMMARY:
Aging is associated with a decline in muscle mass, strength, and physical function, leading to muscle mass loss and weakness. These concerns can impact an individual's functional independence and quality of life (QOL). Dietary protein stimulates muscle protein growth. Current studies suggest that optimal protein intake for older adults is greater than the Recommended Dietary Allowance. Barriers to consuming protein-rich foods in older adults include reductions in taste and smell, dentition, dexterity, and changes in living situation. Therefore, nutritional interventions are needed to effectively improve eating behaviors, diet quality, and stimulate muscle growth and strength. These interventions will help prevent, manage, and promote muscle mass loss recovery. Older adults may not be aware of their changing nutrient needs and therefore may lack the skills to prepare nutritionally adequate foods properly. Cooking demonstrations, or culinary medicine (CM), can help teach healthy cooking to reduce potential red meat consumption barriers and improve community-dwelling older adults' dietary habits. Thus, CM can be a novel strategy to improve diet quality in older adults and promote and augment at-home cooking. CM is an evidenced-base field that combines skills of preparing, cooking, and presenting food with the science of medicine. This field can help to accomplish potential eating behaviors and health outcome improvements. A tailored CM program can be an effective strategy that could reduce barriers in protein intake that will enable older adults to age well and productively.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* physically active
* able to cook for oneself
* willing to complete two blood draws

Exclusion Criteria:

* <65 years old
* sedentary lifestyle
* bleeding disorder
* heart pacemaker
* type 1 diabetics and type 2 diabetics taking insulin
* current smokers
* amputees

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Dual Energy X-ray Absorptiometry (DXA) | Baseline and change from baseline muscle mass and fat mass at 4 months
  DXA will measure full body muscle mass and fat mass in grams.

SECONDARY OUTCOMES:
Protein questionnaire | Baseline and through study completion, an average of 4 months
  The subject will fill out an online modified version of the rapid self-administered dietary protein food frequency questionnaire. This questionnaire contains 20-items evaluating the weekly intake of different types of meat, dairy, eggs, beans to provide the weekly protein intake in grams.
Cooking Effectiveness Questionnaire | Baseline and through study completion, an average of 4 months
  Questionnaire to record effectiveness of culinary medicine cooking videos based on a scale of from "completely confident" to "not confident at all"
Body mass index in kg/m^2 | Baseline and change from baseline BMI at 4 months
  Weight in kg and height in meters will be used to calculate BMI
Weight in lbs | Baseline and change from baseline weight at 4 months
  Weight will be measure to the nearest 0.1 lbs
Height in inches | Baseline
  Height will be measured to the nearest 0.1 in using a stadiometer.
Steps | through study completion, an average of 4 months
  Subjects will be provided a Garmin Vivofit 4 watch to monitor their steps throughout the study
Grip strength | Baseline and change from baseline grip strength at 4 months
  Grip strength will be measured by a handheld dynamometer. The subject will be asked to used the handheld dynamometer three times for each to obtain the average of the three test results.
Physical activity questionnaire | Baseline and change from baseline CHAMPS at 4 months
  Community Healthy Activities Model Program for Seniors (CHAMPS) is 41-items that assess the weekly frequency and duration of various physical activities typically undertaken by older adults. Each question ask how many times a week the participant partake in the activity then ask how many total hours a week the participant did the activity. The frequency per week of all exercise-related activities were calculated by the sum frequency scores/week for each of the activities. The higher the score, the better the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Salas-Groves E, Alcorn M, Childress A, Galyean S. The Effect of Web-Based Culinary Medicine to Enhance Protein Intake on Muscle Quality in Older Adults: Randomized Controlled Trial. JMIR Form Res. 2024 Feb 13;8:e49322. doi: 10.2196/49322. PMID 38349721